CLINICAL TRIAL: NCT00094679
Title: A Randomized Trial Comparing Part-time Versus Minimal-time Patching for Moderate Amblyopia
Brief Title: Trial Comparing Part-time Versus Minimal-time Patching for Moderate Amblyopia
Acronym: ATS2B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Roy W. Beck, M.D., Ph.D., Jaeb Center for Health Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATS2B; 2U10EY011751 (NIH)
Record Dates: First submitted 2004-10-21; First posted 2004-10-22 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2hrs daily patching (Active Comparator): 2 hours patching per day to cover the sound eye
  Interventions: Device: Eye patch
- 6hrs daily patching (Active Comparator): 6 hours per day patching to cover the sound eye
  Interventions: Device: Eye patch

INTERVENTIONS:
Device: Eye patch — adhesive patch to cover the sound eye
  Other Names: Coverlet; Opticlude

SUMMARY:
The goals of this study are:

* To determine whether the visual acuity improvement obtained with part-time (6 hours) patching is equivalent to the visual acuity improvement obtained with minimal patching (2 hours) for moderate amblyopia.
* To develop more precise estimates than currently available for the visual acuity improvement that occurs during treatment of amblyopia with patching.
* To identify factors that may be associated with successful treatment of amblyopia with patching.

DETAILED DESCRIPTION:
Amblyopia is the most common cause of monocular visual impairment in both children and young and middle-aged adults. Patching has been the mainstay of amblyopia therapy. It is generally held that the response to treatment is best when it is instituted at an early age, particularly by age two or three, and is poor when attempted after eight years of age.

For moderate amblyopia, patching is the most commonly prescribed treatment although other modalities such as atropine penalization are also prescribed. There is no specific patching regimen that is widely accepted for treatment of moderate amblyopia and limited or no data available to favor the use of one specific regimen; both minimal occlusion (e.g., 2 hours per day) and six or more hours per day of patching are prescribed in clinical practice.

The study is a randomized trial comparing daily patching regimes for children with moderate amblyopia. It will consist of about 160 children. Patients in the moderate (20/40-20/80) group will patch part-time (6 hours) or minimal time (2 hours) of each day for the 4-month study period. There are at least two follow up visits during the 4-month period. Visual acuity is the major study outcome. It is assessed at the 4-month exam.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be less than 7 years of age with the original cause of amblyopia as strabismus or anisometropia.
* Visual Acuity in the amblyopic eye must be between 20/40 and 20/80.
* Visual acuity in the sound eye of 20/40 or better.
* There must be at least 3 lines of acuity difference between the two eyes.

Exclusion Criteria:

* Patching treatment (other than spectacles) within six months prior to enrollment and other amblyopia treatment of any type used within one month prior to enrollment.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 189 (Actual)
Dates: Start 2001-05; Primary Completion 2002-07 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Visual acuity improvement | 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael X Repka, M.D., Study Chair — Wilmer Eye Institute
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States

REFERENCES:
- [Background] Repka MX, Beck RW, Holmes JM, Birch EE, Chandler DL, Cotter SA, Hertle RW, Kraker RT, Moke PS, Quinn GE, Scheiman MM; Pediatric Eye Disease Investigator Group. A randomized trial of patching regimens for treatment of moderate amblyopia in children. Arch Ophthalmol. 2003 May;121(5):603-11. doi: 10.1001/archopht.121.5.603. PMID 12742836
- [Derived] Repka M, Simons K, Kraker R; Pediatric Eye Disease Investigator Group. Laterality of amblyopia. Am J Ophthalmol. 2010 Aug;150(2):270-4. doi: 10.1016/j.ajo.2010.01.040. Epub 2010 May 8. PMID 20451898